CLINICAL TRIAL: NCT06389955
Title: A Phase 1, Randomized, Study in Healthy Volunteers to Assess Relative Bioavailability and Effect of Food on Capsule and Tablet Formulations of TP-3654
Brief Title: Assessment of Relative Bioavailability and Effect of Food on Capsule and Tablet Formulations of TP-3654
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TP-3654-103
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — TP 3654

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part A - Sequence 1 (Experimental): Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants randomly assigned to Sequence 1 will take TP 3654 with or without food as follows: Day 1 - 480mg (4 x 120mg capsules) once daily with low fat meal, Day 4 - 480mg (4 x 120mg capsules) once daily fasted, Day 7 - 480mg (4 x 120mg capsules) once daily with high fat meal, and Day 10 - 480mg (2 x 240mg tablets) once daily fasted.
  Interventions: Drug: TP 3654
- Part A - Sequence 2 (Experimental): Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants randomly assigned to Sequence 2 will take TP 3654 with or without food as follows: Day 1 - 480mg (4 x 120mg capsules) once daily fasted, Day 4 - 480mg (2 x 240mg tablets) once daily fasted, Day 7 - 480mg (4 x 120mg capsules) once daily with low fat meal, and Day 10 - 480mg (4 x 120mg capsules) once daily with high fat meal.
  Interventions: Drug: TP 3654
- Part A - Sequence 3 (Experimental): Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants randomly assigned to Sequence 3 will take TP 3654 with or without food as follows: Day 1 - 480mg (2 x 240mg tablets) once daily fasted, Day 4 - 480mg (4 x 120mg capsules) once daily with high fat meal, Day 7 - 480mg (4 x 120mg capsules) once daily fasted, and Day 10 - 480mg (4 x 120mg capsules) once daily with low fat meal.
  Interventions: Drug: TP 3654
- Part A - Sequence 4 (Experimental): Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants randomly assigned to Sequence 4 will take TP 3654 with or without food as follows: Day 1 - 480mg (4 x 120mg capsules) once daily with high fat meal, Day 4 - 480mg (4 x 120mg capsules) once daily with low fat meal, Day 7 - 480mg (2 x 240mg tablets) once daily fasted, and Day 10 - 480mg (4 x 120mg capsules) once daily fasted.
  Interventions: Drug: TP 3654
- Part B - Sequence 1 (Experimental): Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants randomly assigned to Sequence 1 will take TP 3654 tablets with or without food as follows: Day 1 - 480mg once daily with low fat meal, Day 4 - 480mg once daily fasted, and Day 7 - 480mg once daily with high fat meal.
  Interventions: Drug: TP 3654
- Part B - Sequence 2 (Experimental): Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants randomly assigned to Sequence 2 will take TP 3654 tablets with or without food as follows: Day 1 - 480mg once daily fasted, Day 4 - 480mg once daily with high fat meal, and Day 7 - 480mg once daily with low fat meal.
  Interventions: Drug: TP 3654
- Part B - Sequence 3 (Experimental): Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants randomly assigned to Sequence 3 will take TP 3654 tablets with or without food as follows: Day 1 - 480mg once daily with high fat meal, Day 4 - 480mg once daily with low fat meal, and Day 7 - 480mg once daily fasted.
  Interventions: Drug: TP 3654

INTERVENTIONS:
Drug: TP 3654 — TP 3654 is an investigational orally delivered drug

SUMMARY:
This study comprised of 2 parts, Part A and Part B. Part B will only be conducted if the relative bioavailability of the tablet formulation was at least 70% of the capsule formulation.

DETAILED DESCRIPTION:
Part A is a randomized, single-dose, 4-period, 4-way cross-over study to evaluate the effect of food on the TP 3654 capsule and assess the relative bioavailability of the TP-3654 capsule versus tablet formulations. Following a screening period of up to 28 days, eligible participants will be admitted to the clinical research unit (CRU) on Day -1. Participants will fast overnight from Day -1 to Day 1. On Day 1, participants will be randomly assigned to a treatment sequence, and they will receive TP-3654 per their assigned sequence.

Part B is a randomized, single-dose, 3-period, 3-way cross-over study to evaluate the effect of food on the PK of the TP-3654 tablet formulation. Following a screening period of up to 28 days, eligible participants will be admitted to the CRU on Day -1. As with Part A, participants will fast overnight from Day -1 to Day 1. On Day 1, they will be randomly assigned to a treatment sequence, and they will receive TP-3654 per their assigned sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent.
2. Participant is ≥ 18 to ≤ 65 years of age.
3. Participant is willing and able to consume the prescribed standard meals.
4. Participant agrees to use an acceptable method of contraception as described in Section 8.5.4 for the duration of the study and agrees to continue use for 3 months after the final dose (male participants) or for 6 months after the final dose (female participants).
5. Male participant agrees not to donate sperm during the study and for 3 months after the last dose of study drug. Female participant agrees not to donate eggs for the duration of the study and for 6 months after the last dose of study drug.
6. Participant has a BMI ≥ 18.5 and ≤ 32 kg/m2 at screening.
7. Participant is generally healthy, as determined by the Investigator based on medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG) at screening. In particular:

   1. Clinical laboratory results must be within normal range
   2. Body temperature is < 38°C (100.3°F).
   3. Blood pressure and heart rate are within normal limits (systolic blood pressure is ≥ 90 to ≤ 150 mmHg; supine diastolic blood pressure is ≥ 50 to ≤ 90 mmHg; heart rate is ≥ 40 to ≤ 90 bpm) at screening.
   4. Average triplicate corrected QT interval (QTcF) ≤ 430 msec (for male participants) or ≤ 450 msec (for female participants).
8. Participant agrees to avoid the use of concomitant medications (except hormonal contraception or medication provided by the site staff under the direction of the Investigator) from screening through the final follow-up visit.
9. Participant agrees to abstain from alcohol, recreational drugs (including marijuana), and nicotine from screening through the final follow-up visit.
10. Participant is willing and able to remain confined in the Clinical Research Unit for the duration of the inpatient period (13 days for Part A or 10 days for Part B)

Exclusion Criteria:

1. Participant is pregnant (as evidenced by a positive pregnancy test) or nursing.
2. Participant reports a history (within 3 years prior to screening) of any clinically significant neurological, gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, endocrine, hematological, dermatological, psychological, or other disorders as determined by the Investigator.
3. Participant reports use of CYP3A hepatic microsomal enzyme interacting drugs (such as voriconazole, fluconazole, cimetidine) within 30 days prior to admission.
4. Participant reports being exposed to an investigational product (drug, biologic, or device) within 30 days preceding the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).
5. Participant reports having a surgical procedure that may affect drug absorption, distribution, metabolism, and/or excretion (eg, bariatric procedure, cholecystectomy). Appendectomy is acceptable.
6. Participant reports donating blood within 8 weeks before the first dose administration.
7. Participant reports a history of alcohol or drug use disorder within 2 years before screening.
8. Participant has a positive drug screening test reflecting use of recreational drugs.
9. Participant reports being a current smoker or use of nicotine products (eg, nicotine gum or patch, vaporized nicotine, chewing tobacco)
10. Participant has poor venous access or has a history of difficulty providing blood samples.
11. Participant reports any condition or has any finding that would, in the Investigator's opinion, put the participant or study conduct at risk if the participant were to be enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Part A - The maximum concentration (Cmax) of TP-3654 in a capsule formulation | 2 weeks
Part A - The area under the curve (AUC) of TP-3654 in a capsule formulation | 2 weeks
Part A - Ratio of Peak Plasma Concentration (Cmax) of TP-3654 tablet versus TP-3654 capsule under fasted conditions | 2 weeks
Part B - The maximum concentration (Cmax) of TP-3654 in a tablet formulation | 2 weeks

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAE) | 6 weeks
  TEAEs will be monitored from first dose to 30 days after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Investigative Site, Secaucus, New Jersey, United States